CLINICAL TRIAL: NCT05068713
Title: High Versus Low Blood-Pressure Target in the Post Operative Care of Liver Transplantation
Brief Title: High Versus Low Blood-Pressure Target in the Post Operative Care of Liver Transplantation A Randomized, Controled, Open and Unicentric Trial.
Acronym: LIVER-PAM
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Sao Paulo General Hospital (Other)
Responsible Party: Principal Investigator, Rodolpho Augusto de Moura Pedro, Principal investigator, University of Sao Paulo General Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: LIVER-PAM
Record Dates: First submitted 2021-09-24; First posted 2021-10-06 (Actual); Last update posted 2024-01-17 (Actual); Status verified 2024-01

CONDITIONS: Liver Transplant; Complications

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hihg Target Mean Arterial Pressure (Experimental): Target of mean arterial pressure of 85-90 mmHg in ther first 24h after liver transplant.
  Interventions: Other: Usual Care + High Target of Mean Arterial Pressure
- Low Target Mean Arterial Pressure (Active Comparator): Target of mean arterial pressure of 65-70 mmHg in ther first 24h after liver transplant.
  Interventions: Other: Usual Care

INTERVENTIONS:
Other: Usual Care + High Target of Mean Arterial Pressure — Targeting the weaning of vasopressors to a mean arterial pressure of 85-90mmHg in the first 24h after liver trasnplant.
  Arms: Hihg Target Mean Arterial Pressure
Other: Usual Care — Targeting the weaning of vasopressors to a mean arterial pressure of 65-70mmHg in the first 24h after liver trasnplant.
  Arms: Low Target Mean Arterial Pressure

SUMMARY:
LIVER PAM

A randomized, controled, open and unicentric trial comparing high (MAP 85-90 mmHg) and low (65-70 mmHg) target of mean arterial pressure in the first 24 hours after liver transplantation.

ELIGIBILITY:
Inclusion Criteria:

* Older than 18 y
* Admitted in the ICU for a post operative care after liver transplant

Exclusion Criteria:

* Consent refusal
* Liver transplant due to acute liver failure
* Renal transplant ( Previous or concomitant)
* Refusal from the healthcare provider responsible for the patient
* Renal substitution therapy in the prior 15 days
* Pregnancy
* Re-Transplant (Liver transplant in the previous 6 month)
* Hepatorenal syndrome current treatment (Use of terlipressin + Albumin)
* Refractory and persistent shock during or after transplant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 174 (Actual)
Dates: Start 2021-08-24 (Actual); Primary Completion 2024-01-05 (Actual); Study Completion 2024-01-05 (Actual)

PRIMARY OUTCOMES:
incidence of Acute Kidney Disfunction | 7 days
  Incidence of acute kidney Disfunction according to kdigo criteria.

SECONDARY OUTCOMES:
Mortality | 28 days
  percentage of mortality in 28 days
re-transplant | 28 days
  percentage of re-transplant in 28 days
Lenght of Hospitay Stay | 28 days
  LOS in 28 days
Lenght of ICU Stay | 28 days
  ICU LOS in 28 days
Days alive and out of hospital in 28 days | 28 days
  Number of days alive and out of hospital in 28 days
Substitutive Renal Therapy | 7 days
  percentage of TSR in 7 days
Days Alive and free of renal disfunction | 28 days
  Days Alive and free of renal disfunction in 28 days
Acute kidney insufficiency according to Urinary NGAL on d0 and D2 | 0d and 2d
  Percentage of renal disfunction according to NGAL criteria on D0 and D2
MAKE28 | 28 days
  Major Kidney Events ( Death, persistent acute kidney disfunction or need of RRT in 28 days)
Liver graft primary disfunction ( Initial Poor Function) | 7 days
  percentage of Initial Poor Function in 7 days
Liver graft primary disfunction (primary nonfunction) | 10 days
  percentage of primary nonfunction in 10 days
Surgical site infection | 28 days
  percentage of SSI in 28 days
Need of Transfusion | 7 days
  percentage of Transfusion requirement in 7 days
Postoperative Major bleeding in 7 days | 7 days
  Bleeding that requires 2 units of blood transfusion in a single day or the need of a reoperation due to bleeding in the first 24 hours after surgery.
Incidence of Arrythmia requiring clinical treatment | 7 days
  percentage of Arrhythmia requiring treatment in 7 days

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Das Clínicas Da Faculdade de Medicina Da Universidade de São Paulo, São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Pedro RAM, Scharranch BC, Araujo LO, Brandao LS, Andrade LDC, Andraus W, D'Albuquerque LAC, Malbouisson LMS. High versus low mean arterial pressure target in liver transplant patients. An open, controlled, single-center, randomized clinical trial - Protocol and methods (LIVER-PAM). Crit Care Sci. 2023 Mar 1;35(1):11-18. doi: 10.5935/2965-2774.20230336-en. PMID 37712725